CLINICAL TRIAL: NCT06657040
Title: Music for Surgical Intensive Care (MUSIC)
Acronym: (MUSIC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 74416523.0.1001.5249
Record Dates: First submitted 2024-09-11; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-07

CONDITIONS: DELIRIUM
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTERVENTION (Active Comparator): The intervention group will receive a soundtrack through individual choice of anti-noise headphones. The music offer platform will be provided by an application developed by MusicCare (www.music.care/en/index.html) in two periods of the day (09:00 and 16:00), lasting 45 minutes each, for up to seven postoperative days or until discharge from the unit (whichever occurs first).
  Interventions: Other: MUSIC
- STANDARD TREATMENT (Placebo Comparator): IN THIS ARM, PATIENTS WILL UNDERGO STANDARD TREATMENT IN THE ICU WHERE THEY ARE ADMITTED AND FOR 45 MINUTES, TWICE A DAY, NOISE-CANCELLING HEADPHONES WILL BE USED WITHOUT PLAYING MUSIC.
  Interventions: Other: MUSIC

INTERVENTIONS:
Other: MUSIC — The intervention group will receive a soundtrack through individual choice of anti-noise headphones. The music offer platform will be provided by an application developed by MusicCare (www.music.care/en/index.html) in two periods of the day (09:00 and 16:00), lasting 45 minutes each, for up to seven postoperative days or until discharge from the unit (whichever occurs first). MusicCare has been widely tested in several countries and there are a large number of publications in anesthesiology, ICU, cardiology and neurology, among other specialties, demonstrating its safety and efficacy69,70. Patients who were hospitalized for more than 48 hours, that is, who received a minimum of 4 intervention periods, will be considered as patients with effective intervention. Patients with less time will be evaluated in the form of intention to treat.

SUMMARY:
Intensive care units (ICUs) are environments specialized in the care of critically ill patients. Despite significant advances, ICUs are often seen as a dehumanized environment. Among the various stressors in ICUs, anxiety, pain, psychomotor agitation and mental confusion, need for mechanical restraint, lack of privacy, noise, restricted visiting time with family members and excessive lighting stand out. The tripod composed of pain, anxiety and delirium (often associated with the presence of psychomotor agitation, mental confusion and altered level of consciousness) has a high incidence and morbidity. A set of prevention, intensity reduction and treatment measures has been proposed for these conditions, with a growing number of scientific evidence supporting their routine use.

Elderly patients tend to be particularly susceptible to the stressors described above. This aspect represents an additional source of concern for ICUs, since the elderly today represent the majority of patients admitted to ICUs. Hospitalization in ICUs after surgical procedures is often an unknown moment for the individual and, consequently, associated with the development of numerous unpleasant sensations, directly interfering with the patient's recovery.

Music as a therapy tool in medical practice has been used since 1890. After a little more than two decades, in 1914 it was applied in a surgical procedure by physician Evan Kane as a way of "calming patients and diverting attention from fear". associated with combined therapy with local anesthesia. In this context, being a low-cost tool, with minimal adverse effects and high acceptability, the use of music has proven to be a great ally in the arsenal of non-pharmacological therapies for the prevention of delirium, anxiety and pain.

We intend, through a randomized multicenter clinical trial, to investigate whether the use of music as therapy is capable of reducing the incidence of anxiety, pain and delirium in elderly patients undergoing surgical procedures and hospitalized during the postoperative period in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery admitted to the ICU in the immediate period after the surgical procedure; · Age equal to or greater than 65 years

Exclusion Criteria:

* · Moderate to severe dementia, defined by 2 to 3 points in the clinical dementia rating (CDR)66;

  * Impossibility of verbal communication (eg: aphasia);
  * Lack of understanding of the Portuguese language;
  * Inability to listen to music due to hearing impairment or intolerance to the use of headphones;
  * Mechanical ventilation for more than 12 hours;
  * Richmond Agitation Sedation Scale (RASS) less than or equal to 324;
  * Neurosurgical and craniofacial procedures;
  * Refusal or failure to sign the free and informed consent form (TCLE).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
combined frequency of delirium and anxiety | SEVEN DAYS
  The primary endpoint is the combined frequency of delirium and anxiety during the first 7 days of ICU stay Assessments will be performed using the form developed for the study, consisting of the CAM-ICU 7, the numeric pain scale (NRS) and the HADS-A scale. Additionally, the form will document the vital signs: systolic blood pressure, diastolic blood pressure and heart rate measured immediately before and after the intervention in the two periods of the day, in addition to data referring to the presence of pain and episodes of psychomotor agitation and/or delirium, as well as the use of analgesics and opioids in the period referring to the 12 hours prior to the application of the intervention. The CAM-ICU7 and NRS tools will be applied twice a day before and after the intervention, as well as the measurement of vital signs, while the HADS-A scale will be applied only once a day in the morning assessment.

IPD SHARING:
Plan to Share IPD: No